CLINICAL TRIAL: NCT07319650
Title: Efficacy Of Platelet Rich Fibrin (PRF) In Neurosensory Disturbance Among Patients With Mandibular Body Fractures
Acronym: PRF NSD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Health Sciences Lahore (Other)
Responsible Party: Principal Investigator, Muhammad umair shakir, Postgraduate Resident (MDS) Oral & Maxillofacial Surgery, University of Health Sciences Lahore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ERB172/ 2 /10-10-2024/S1 ERB
Record Dates: First submitted 2025-12-20; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Neurosensory Disturbance; Mandibular Body Fractures
Keywords: Neurosensory Disturbance; Platelet Rich Fibrin; Mandibular body fractures

STUDY DESIGN:
Intervention Model Description: Experimental Group= The group in which PRF will be placed over mental nerve during open reduction and internal fixation of patients with mandibular body fractures.
  Control Group= The group in which PRF will not be placed over mental nerve during open reduction and internal fixation of patients with mandibular body fractures.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Case Group (Experimental): The group in which PRF will be placed over mental nerve during open reduction and internal fixation of patients with mandibular body fractures involving mental foramen.
  Interventions: Other: Platelets rich Fibrin
- Control Group (No Intervention): The group in which PRF will not be placed over mental nerve during open reduction and internal fixation of patients with mandibular body fractures.

INTERVENTIONS:
Other: Platelets rich Fibrin — PRF is the second generation autologous platelet concentrate that is obtained from patient's own blood in simple and cost effective manner. PRF is comprised of three main specifications. First, the existence of platelets and their active growth factors i.e. platelet derived growth factor (PDGF), vascular endothelial growth factor (VEGF), transforming growth factor (TGF), insulin-like growth factor (IGF) and epidermal growth factor (EGF). Second, the role of leukocytes and cytokines i.e. TNF alpha, IL-6 and IL-1ɓ in anti-inflammatory response and immune modulation. Third, the fibrin meshwork where these platelets, cytokines and growth factors are embedded and subsequently released after a short period
  Other Names: PRF
  Arms: Case Group

SUMMARY:
Mandibular body fractures frequently result in inferior alveolar nerve (IAN) and mental nerve injuries which ultimately leads to paresthesia of chin and lower lip area. The objective of this study is to evaluate the efficacy of platelet rich fibrin (PRF) application to mental nerve during open reduction and internal fixation (ORIF) of patients having neurosensory disturbance (NSD) following mandibular body fracture involving mental foramen. The PRF application to mental nerve in mandibular body fractures will not only aid in hard and soft tissue healing but also prove to be a game changer for a holistic healing of a patient rather than separate surgical procedures for nerve repair such as microsurgery, grafting, tissue glues, laser.

Alternate Hypothesis HA= The application of PRF to the mental nerve during open reduction and internal fixation of mandibular body fractures involving the mental foramen significantly improves neurosensory recovery compared to cases where PRF is not applied.

Null Hypothesis HO= The application of PRF to the mental nerve during open reduction and internal fixation of mandibular body fractures involving the mental foramen does not significantly improve neurosensory recovery compared to cases where PRF is not applied.

DETAILED DESCRIPTION:
Oral and Maxillofacial surgical procedures such as maxillofacial trauma treatments,TMJ surgeries, cyst enucleation, tumor resection, orthognathic surgeries may result in nerve injuries. Bilateral sagittal split osteotomy can result in damage to IAN nerve. Mandibular fractures can result in damage to IAN/ mental nerve as result of trauma. The frequency of temporary IAN injury is 0.5-5%, whereas permanent injury is <1% and can result in numbness or paresthesia in lower lip and chin area .

The use of PRF may provide a beneficial effect in virtue because it contains several growth factors and may enhance epineurium fibroblast regeneration. PRF has better efficacy than PRP and normal saline (control) in functional nerve recovery (Khojasteh et al.,2016). The use of PRF placement in mandibular body fractures will not only aid in hard and soft tissue healing but also prove to be a game changer for a holistic healing of a patient (Preponement et al.,2013) rather than separate surgical procedures for nerve repair such as microsurgery, grafting, tissue glues, laser.

Limited studies have been done regarding the role of PRF in neurosensory disturbance following mandibular body fractures. The most recent study conducted by Tabrizi et al.(2024) who studied the role of PRF in neurosensory recovery following mandibular body fractures. In this study PRF was placed on IAN between fracture segments. This study had several limitations such as low sample size and there was no direct application of PRF to mental nerve, which may be a factor in NSD. The actual sample size was lower i.e 25 patients as compared to their calculated sample size i.e 30, because 5 patients did not return for follow-up. Our study will provide more significant data related to efficacy of PRF application to mental nerve in patients having neurosensory disturbance following mandibular body fracture involving mental foramen. The PRF application to mental nerve in mandibular body fractures will not only aid in hard and soft tissue healing but also prove to be a game changer for a holistic healing of a patient rather than separate surgical procedures for nerve repair such as microsurgery, grafting, tissue glues, laser.

ELIGIBILITY:
Inclusion Criteria:

* Patients having neurosensory disturbance following mandibular body fracture involving mental foramen and pre-operative TPD discrimination score '0' or '1' will be selected in this study ( as per operational definition). TPD discrimination will be recorded; Preoperatively Immediately post operatively After 6 months

Age 15-40years, Both Gender ASA_1

Exclusion Criteria:

* Comminuted mandibular fractures Previously treated cases of fractures Patients with history of neurological disorders Comorbid patients

Ages: 15 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Neurosensory Recovery | Patients having NSD following mandibular body fractures involving mental foramen and pre-operative TPD discrimination score '0' or '1' will be selected in this study .TPD discrimination will be recorded; Preoperatively Immediately After six months
  Neurosensory disturbance in patients following mandibular body fractures involving mental foramen will be assessed using Two-point discrimination as the primary variable. TPD will be recorded as the minimum distance between two pinpricks that patient could recognize at lower lip and chin area. TPD will be performed by placing a sliding caliper on the skin of chin and mucosa of lower lip. Following scoring criteria has been used in literature (khojasteh et al.,2016).
  TPD >20mm = Score 0 14-20mm= Score 1 <14mm= Score 2

CONTACTS AND LOCATIONS:
Overall Officials: Dr Gulraiz Zulfiqar, FCPS(OMFS), Study Director — Associate professor and Head of Department Oral & Maxillofacial Surgery, Allama Iqbal Medical College/ Jinnah Hospital Lahore
Locations (1):
- Allama Iqbal Medical College/ Jinnah Hospital Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Yadav S, Sachdeva A, Verma A.2011. Inferior alveolar nerve damage following removal of mandibular third molar teeth. Journal of Innovative Dentistry, 1:1-4.
- [Background] Wu CL, Lee SS, Tsai CH, Lu KH, Zhao JH, Chang YC. Platelet-rich fibrin increases cell attachment, proliferation and collagen-related protein expression of human osteoblasts. Aust Dent J. 2012 Jun;57(2):207-12. doi: 10.1111/j.1834-7819.2012.01686.x. PMID 22624763
- [Background] Thurmüller P, Dodson TB, Kaban LB.2001. Nerve injuries associated with facial trauma: natural history, management, and outcomes of repair. Oral Maxillofac Surg Clin,13:283-293.
- [Background] SUNDERLAND S. A classification of peripheral nerve injuries producing loss of function. Brain. 1951 Dec;74(4):491-516. doi: 10.1093/brain/74.4.491. No abstract available. PMID 14895767
- [Background] Reza Tabrizi, DMD1, Hamidreza Moslemi, DMD2, Shervin Shafiei, DMD1,Ramtin Dastgir, DDS3 and Zachary S. Peacock, DMD, MD.2024.FACS4Craniomaxillofacial Trauma &Reconstruction , Vol. 0(0) 1-7
- [Background] Tabrizi R, Pourdanesh F, Jafari S, Behnia P. Can platelet-rich fibrin accelerate neurosensory recovery following sagittal split osteotomy? A double-blind, split-mouth, randomized clinical trial. Int J Oral Maxillofac Surg. 2018 Aug;47(8):1011-1014. doi: 10.1016/j.ijom.2018.04.010. Epub 2018 May 4. PMID 30954205
- [Background] Padmaraj Hegde, Bhadrinath Sai Swaroop, Tripthi Shetty.2021.Department of Oral and Maxillofacial Surgery, NITTE University, AB Shetty Memorial Institute of Dental Sciences 575018, Mangalore, INDIA Nat. Volatiles & Essent. Oils,8(5):10566-10571
- [Background] Libersa P, Savignat M, Tonnel A. Neurosensory disturbances of the inferior alveolar nerve: a retrospective study of complaints in a 10-year period. J Oral Maxillofac Surg. 2007 Aug;65(8):1486-9. doi: 10.1016/j.joms.2007.03.023. PMID 17656272
- [Background] Khojasteh A, Hosseinpour S, Nazeman P, Dehghan MM. The effect of a platelet-rich fibrin conduit on neurosensory recovery following inferior alveolar nerve lateralization: a preliminary clinical study. Int J Oral Maxillofac Surg. 2016 Oct;45(10):1303-8. doi: 10.1016/j.ijom.2016.06.003. Epub 2016 Jun 30. PMID 27371997
- [Background] Boffano P, Roccia F, Gallesio C, Karagozoglu K, Forouzanfar T. Inferior alveolar nerve injuries associated with mandibular fractures at risk: a two-center retrospective study. Craniomaxillofac Trauma Reconstr. 2014 Dec;7(4):280-3. doi: 10.1055/s-0034-1375169. Epub 2014 Jun 5. PMID 25383147
- [Background] Abhinav RP, Selvarasu K, Maheswari GU, Taltia AA. The Patterns and Etiology of Maxillofacial Trauma in South India. Ann Maxillofac Surg. 2019 Jan-Jun;9(1):114-117. doi: 10.4103/ams.ams_233_18. PMID 31293938